CLINICAL TRIAL: NCT02868333
Title: Determinants of Health Status and Quality of Life in Patients With Primary Immunodeficiencies Inhereted Diagnosed During Childhood
Acronym: CEREDIH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-10; 2012-A00338-35 (Other: ANSM)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Primary Immune Deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Most children with primary immune deficiency (PID) now reach adulthood. However, few studies have evaluated their health status and health related quality of life (HRQoL).

Objective: To investigate long-term morbidity, the French Reference Center for PIDs initiated a prospective multicenter cohort: the F-CILC (French Childhood Immune deficiency Long-term Cohort). The data collected will be used to assess the physical health condition of patients who reached adulthood and the impact on their quality of life.

Methods: Patients are asked to complete health status questionnaires. A severity score (grade1 ["mild"] to grade 4 ["life-threatening"]) is assigned to each health condition. The HRQoL of patients is compared to age- and sex-matched French normal values using the SF36 HRQoL questionnaire.

Capsule summary. This will be the first study of adult survivors of childhood PID describing how the burden of health conditions affect their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary immune deficiency diagnosed during childhood

Exclusion Criteria:

* Patients not willing to answer to quality of life questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with primary immune deficiency diagnosed during childhood and followed in refereries center for this desease
Sampling Method: Non-Probability Sample
Enrollment: 1780 (Actual)
Dates: Start 2012-05; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Numbers of patient with PID diagnosed during childhood experiencing a heavy burden of health conditions affecting their quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Vincent BARLOGIS, MD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barlogis V, Mahlaoui N, Auquier P, Fouyssac F, Pellier I, Vercasson C, Allouche M, De Azevedo CB, Moshous D, Neven B, Pasquet M, Jeziorski E, Aladjidi N, Thomas C, Gandemer V, Mazingue F, Picard C, Blanche S, Michel G, Fischer A. Burden of Poor Health Conditions and Quality of Life in 656 Children with Primary Immunodeficiency. J Pediatr. 2018 Mar;194:211-217.e5. doi: 10.1016/j.jpeds.2017.10.029. Epub 2017 Dec 6. PMID 29198545